CLINICAL TRIAL: NCT05170607
Title: Investigation of Specific Biomarkers in Patients With Atrial Fibrillation Who Undergo Interventional Treatment
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Responsible Party: Sponsor
Other Study IDs: 121122200154-7
Record Dates: First submitted 2021-12-24; First posted 2021-12-28 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; protein microarray; proteomic biomarkers; PV dependent atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PV associated atrial fibrillation
  Interventions: Diagnostic Test: Proteomic analysis by antibody microarrays
- non-PV associated arrhythmic focuses
  Interventions: Diagnostic Test: Proteomic analysis by antibody microarrays
- Healthy volunteers
  Interventions: Diagnostic Test: Proteomic analysis by antibody microarrays

INTERVENTIONS:
Diagnostic Test: Proteomic analysis by antibody microarrays — Proteomic analysis by antibody microarrays can be used to identify novel biomarkers and to investigate various signaling pathways including protein phosphorylation and protein-protein interactions. Microchips are manufactured as a matrix of a number of immobilized antibodies covalently bound to the glass, membrane, or gel surfaces. Microchips are used for serum proteomic studies in patients with cardiovascular diseases and cancer

SUMMARY:
The two main mechanisms for atrial fibrillation (AF) recurrence after cryoablation include Pulmonary vein (PV) reconnection and the presence of non-PV associated arrhythmic focuses. The aim of this study is to reveal the specific biomarkers by antibody microarrays.

DETAILED DESCRIPTION:
One hundred twenty patients with atrial fibrillation will participate in the study.

They will be divided into three groups.

1. Patients with AF recurrence after the first procedure but with isolated pulmonary veins at the beginning of the second AF ablation b)patients with AF recurrence after repeat PV ablation.
2. Patients with PV-associated atrial fibrillation. The group will be included patients with freedom of atrial fibrillation after PV isolation (first or repeat procedure).
3. Healthy volunteers

Groups would be formed from patients who previously underwent atrial fibrillation ablations and whose blood samples have been taken and placed in a biobank before interventional treatment. The first step will include proteomic serum profiling using antibody microarrays in ten subjects will be split into 3 groups. The second step will include validation of selected protein biomarkers, in the total cohort (N=120).

ELIGIBILITY:
Inclusion Criteria:

• Patient with paroxysmal/persistent atrial fibrillation who underwent interventional treatment

Exclusion Criteria:

* permanent AF
* contraindications to oral anticoagulation or heparin
* chronic kidney disease requiring dialysis
* untreated hypo- or hyperthyroidism
* breast feeding
* pregnancy
* chronic kidney disease requiring dialysis
* decompensated heart failure
* stroke within the last 3 months
* myocardial infarction within the last 3 months
* Percutaneous coronary intervention or Coronary Artery Bypass Grafting within the last 3 months
* active myocarditis
* artificial valve replacement surgery
* severe mitral or aortic stenosis
* coronary artery disease requiring revascularization
* heart transplant

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients 18-85 years old with s paroxismal or persistant atrial fibrillation and prior interventional treatment
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
proteins after validation | 1 year
  number of protein which will be specific for non-PV associated arrhythmic focuses group after validation

SECONDARY OUTCOMES:
proteins after screening | 1 year
  number of protein which will be specific for non-PV associated arrhythmic focuses group after screening

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Center for Preventive Medicine, Moscow, Russia